CLINICAL TRIAL: NCT03608878
Title: Randomized, Controlled, Open Label, Clinical Trial for Adagloxad Simolenin/OBI-821 in Combination With TACE Therapy in Hepatocellular Carcinoma Patients With GALNT14-rs9679162-non-TT Genotype
Brief Title: Adagloxad Simolenin/OBI-821 in Combination With TACE Therapy in HCC Patients With GALNT14-rs9679162-non-TT Genotype
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The biopsies in the first 5 screened patients were all negative for Globo-H, of which positive is required to include the patients.
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chau-ting, Yeh, Director, Liver Research Center; Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGMH/TMUH/VGH-OBI822-HCC001
Record Dates: First submitted 2018-07-23; First posted 2018-08-01 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE alone arm (Active Comparator): TACE (Transarterial Chemoembolization)
  Interventions: Procedure: TACE
- adagloxad simolenin arm (Experimental): TACE plus adagloxad simolenin/OBI-821 adjuvant therapy
  Interventions: Biological: adagloxad simolenin/OBI-821; Procedure: TACE

INTERVENTIONS:
Biological: adagloxad simolenin/OBI-821 — Adagloxad simolenin (OBI-822) is a glyco-conjugated protein comprised of a carbohydrate tumor antigen. Globo H allyl glycoside is covalently linked to a carrier protein KLH, presented in a dominant trimer form with molecular weight between 1200-1395 kDa., to form Adagloxad simolenin (OBI-822) (Globo H-KLH) OBI-821 is a saponin based adjuvant structurally similar to descriptions found in the literature for another adjuvant, QS-21.
  Adagloxad simolenin will be mixed with OBI-821 before administration.
  Arms: adagloxad simolenin arm
Procedure: TACE — Transarterial chemoembolization

SUMMARY:
TACE against HCC is the standard of care for BCLC stage B patients. In this exploratory study, the investigators assess the efficacy of TACE with or without adagloxad simolenin/OBI-821 treatment in GALNT14 "non-TT" HCC population.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common solid cancers worldwide and the third leading cause of cancer-related death. Early stage HCC can be cured by surgical removal or non-surgical ablation procedures, albeit a high recurrence rate up to 75% in 5 years remains an unsolved problem. On the other hand, in patients with unresectable HCC, the "standard therapy" is still under intensive clinical investigations. In patients without portal vein occlusion/thrombosis or extrahepatic metastasis, namely Barcelona Clinical Liver Cancer (BCLC) Stage B, transcatheter arterial chemoembolization (TACE) is believed to be an effective palliative treatment. The beneficial effect of TACE on overall survival has been mild to moderate as reviewed in a previous study. Thus, TACE is generally considered a "palliative" therapy. TACE induces tumor necrosis but at the same time, it also induces angiogenesis owing to the increases of hypoxia-inducible factors and endothelial growth factors to trigger regrowth of tumors.

It has been known that GALNT14 genotype is associated with treatment responses. Patients with GALNT14 "TT" genotype response well to both TACE and chemotherapy.

A new immunotherapy is directed against Globo H, a carbohydrate antigen that is expressed at high levels on the surface of a variety of tumor cells. These Globo H-specific antibodies can effectively induce complement dependent cytotoxicity (CDC) as well as antibody-dependent cell-mediated cytotoxicity (ADCC) by IgM and IgG, respectively, together with other cellular immune responses to kill tumors. In the clinical setting, Globo H has been evaluated as the target of active immunotherapy in a few clinical trials including an ongoing Phase II/III trial of adagloxad simolenin/OBI-821 sponsored by OBI Pharma, Inc., as a potential treatment for stage IV metastatic breast cancers and possibly other cancer types expressing Globo series TACAs. Although vaccination with adagloxad simolenin/OBI-821 did not improve progression-free survival (PFS) in patients with previously treated metastatic breast cancer, in a post-hoc analysis, patients who developed a humoral immune response to Globo H had a longer PFS than those who did not, indicating that adagloxad simolenin/OBI-821 treatment could be of benefit when an antibody response can be developed.

Furthermore, overexpression of tumor-specific antigen Globo H can contribute to enhanced tumor angiogenesis and tumor-associated immune suppression, and in turn, positively correlate with tumor aggressiveness and poor survival in patients. In the present study, only "non-TT" (less favorable) groups will be enrolled and the patients will be randomized to examine the hypothesis that the TACE + adagloxad simolenin/OBI-821 treatment is beneficial in the BCLC class B, advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed Diagnosis of HCC
2. Has a Globo-H or SSEA-3 positive tumor as determined by IHC
3. Never received TACE/ chemotherapy/ radiotherapy or targeted agents prior to this study.
4. Patients should be in BCLC clinical stage B (multinodular asymptomatic tumors without extra-hepatic spread or portal vein invasion) with or without unilateral secondary or tertiary branches of portal vein invasion.
5. Child-Pugh functional class A or B.
6. GALNT14- rs9679162 "non TT" genotype
7. At least 1 measurable lesion must be present.
8. ECOG performance status 0 to 1.
9. Age > 20 years
10. Both men and women enrolled in this trial must use adequate birth control measures during the course of the trial and 4 weeks after last treatment
11. Informed consent must be obtained prior to perform any study procedure.
12. Total bilirubin < 3.0 mg/dL with no evidence of biliary tract obstruction.
13. Appropriate Serum alanine aminotransferase, aspartate aminotransferase, Absolute neutrophil count, Platelets and Serum creatinine

(16) Antiviral treatment for hepatitis B or C is allowed except for interferon.

Exclusion Criteria:

1. BCLC stage A.
2. Presence of extrahepatic metastasis or main portal vein thrombosis.
3. Child-Pugh score = C.
4. Significant cardiac disease as determined by investigator.
5. Serious bacterial infection requiring systemic antibiotics.
6. Pregnancy
7. Expected non-compliance.
8. Uncontrolled illness including, but not limited to, ongoing infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness.
9. Bleeding esophageal or gastric varices within three months without ligation or sclerosis injection therapy.
10. Subjects with known HIV infection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
time-to-ITTVP | From enrollment till 36 months of follow-up.
  time-to-intrahepatic total tumor volume progression

CONTACTS AND LOCATIONS:
Overall Officials: Chau-Ting Yeh, MD, Principal Investigator — LinKou Chang Gung Menorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No